CLINICAL TRIAL: NCT07247357
Title: A Phase 1, Open-Label Study of the Pharmacokinetics of LY4064809 in Healthy Adult Chinese Participants
Brief Title: A Study of LY4064809 in Healthy Adult Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Scorpion Therapeutics, a wholly owned subsidiary of Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 27745; J6M-MC-JSGE (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LY4064809 (Experimental): LY4064809 administered orally
  Interventions: Drug: LY4064809

INTERVENTIONS:
Drug: LY4064809 — administered orally

SUMMARY:
The main purpose of this study is to measure how much LY4064809 gets into the bloodstream and how long it takes the body to eliminate it in healthy participants. It also looks at safety and tolerability in healthy participants. The study drug will be administered orally. The study will last approximately 21 days, excluding screening.

ELIGIBILITY:
Inclusion Criteria:

* Are native Chinese. To qualify as a native Chinese for the purpose of this study, all 4 of the participant's biological grandparents must be of exclusive Chinese descent and born in China
* Are overtly healthy as determined by medical evaluation, including medical history, physical examination, vital signs, and electrocardiogram (ECG) at screening and admission
* Have clinical laboratory test results within the normal range for the population or investigative site, or with abnormalities deemed not clinically significant by the investigator at screening
* Have a body mass index within the range 18 to 32 kilogram per square meter (kg/m²)

Exclusion Criteria:

* History or presence of any of the following conditions, deemed clinically significant by the investigator (or designee), which may significantly alter the absorption, metabolism, or elimination of drugs, constitute a risk when taking the study intervention, or interfere with the data interpretation:

  * metabolic disease, including congenital non-hemolytic hyperbilirubinemia, for example, Gilbert syndrome
  * bile duct disease, including removal of the gall bladder
  * digestive system disease
  * blood disease
  * disease of the nervous system
  * significant history of, or presence of, liver disease, including any abnormal liver function tests, as defined by aspartate aminotransferase, alanine transaminase, or transducin beta-like above the 1.5× upper limit of normal range per the laboratory's reference ranges at screening, or
  * clinically significant, active cardiovascular disease or history of heart attack within 6 months prior to the planned start of LY4064809
* Have a 12-lead ECG abnormality at screening or admission
* History of a major surgical procedure within 30 days prior to screening
* Diagnosed or treated cancer within 5 years prior to screening
* Have known allergies to LY4064809 or related compounds

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2025-10-24 (Actual); Primary Completion 2025-12-16 (Actual); Study Completion 2025-12-16 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY4064809 | Predose on Day 1 Through Day 14
  PK: Cmax of LY4064809
PK: Area Under the Concentration Versus Time Curve (AUC) of LY4064809 | Predose on Day 1 Through Day 14
  PK: AUC of LY4064809

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No